CLINICAL TRIAL: NCT03890692
Title: Assesment of Adenoid Size by Flexible Nasoendoscopy and Lateral Neck Radiography and Its Relation to Clinical Symptoms
Brief Title: Methods of Assessment of Adenoid Size
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ghada mohamed, resident doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOAS
Record Dates: First submitted 2019-03-17; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Adenoid Hypertrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients will undergo flexible nasoendoscopy (Experimental): Endoscopy will be performed by passing the endoscope along either the floor of the nose or just under the middle turbinate. the condition of the nasal mucosa\ septum\ turbinates and the presence of discharge The postnasal space will be assessed . All abnormalities will be recorded .the images will be recorded and assessed separately by two independent otolaryngologists
  Interventions: Procedure: flexible nasoendoscopy

INTERVENTIONS:
Procedure: flexible nasoendoscopy — nasopharyngeal endoscopy : After washing nasal cavities with a sterile physiologic solution to remove secretions or scabs, and decongesting them with an oxymetazoline solution in the subjects with turbinate hypertrophy,
  * Endoscopy will be performed by passing the endoscope along either the floor of the nose or just under the middle turbinate. the condition of the nasal mucosa\ septum\ turbinates and the presence of discharge The postnasal space will be assessed . All abnormalities will be recorded .the images will be recorded and assessed separately by two independent otolaryngologists

SUMMARY:
Chronic nasal obstruction due to adenoid hypertrophy is among the most common health problems affecting children, and adenoidectomy is one of the most common surgical procedures performed in this age group Because of difficulties associated with the use of the objective methods (such as nasopharyngeal endoscopy) in young children, the development of a reliable scale based on the child's symptoms to properly evaluate the need for surgical intervention would be of great value for clinicians. When adenoidectomy is being considered, the diagnosis and documentation of adenoidal hypertrophy become an important issue. Numerous modalities have been used for this task, including trans oral digital palpation and trans oral mirror examination; however, these methods are quite impractical with uncooperative younger children

DETAILED DESCRIPTION:
Assessment of the nasopharynx and adenoids by fibreoptic examination bears the advantage of direct visualization of the postnasal space. In addition, previous studies have demonstrated that adenoid size, as determined by rhinoscopy, was well correlated with clinical symptoms such as nasal obstruction and snoring.

The aim of this study was to compare the effectiveness of lateral neck radiography and video rhinoscopy in assessing adenoid size .

Assessment of the reproducability of these modalities to associated symptoms and, thus, the severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

* children aged 3 _ 14 years old
* clinical diagnosis of adenoid hypertrophy in the form of chronic oral respiration , nasal disorders and snoring
* recurrent otitis media

Exclusion Criteria:

1. patients diagnosed with nasal obstruction due to anatomic malformation ( congenital, choanal atresia, stenosis or septal deviation )
2. age less than 3 years or more than 14 years
3. patient with craniofacial malformation and down syndrome

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
flexible nasoendoscopy in assessment degree of obstruction | baseline
  Endoscopy will be performed by passing the endoscope along either the floor of the nose or just under the middle turbinate. All abnormalities will be recorded. the degree of obstruction will be assesd according to anatomical structures ..such as torus tubarius, vomer, and the soft palate grade 1=none grade 2 reaching torus tubarius, grade 3 reaching torus tubarius and vomer, grade 4 reaching vomer and soft palate.

REFERENCES:
- [Background] Mlynarek A, Tewfik MA, Hagr A, Manoukian JJ, Schloss MD, Tewfik TL, Choi-Rosen J. Lateral neck radiography versus direct video rhinoscopy in assessing adenoid size. J Otolaryngol. 2004 Dec;33(6):360-5. doi: 10.2310/7070.2004.03074. PMID 15971651
- [Background] Talebian S, Sharifzadeh G, Vakili I, Golboie SH. Comparison of adenoid size in lateral radiographic, pathologic, and endoscopic measurements. Electron Physician. 2018 Jun 25;10(6):6935-6941. doi: 10.19082/6935. eCollection 2018 Jun. PMID 30034661
- [Background] Sharifkashani S, Dabirmoghaddam P, Kheirkhah M, Hosseinzadehnik R. A new clinical scoring system for adenoid hypertrophy in children. Iran J Otorhinolaryngol. 2015 Jan;27(78):55-61. PMID 25745612
- [Background] Saedi B, Sadeghi M, Mojtahed M, Mahboubi H. Diagnostic efficacy of different methods in the assessment of adenoid hypertrophy. Am J Otolaryngol. 2011 Mar-Apr;32(2):147-51. doi: 10.1016/j.amjoto.2009.11.003. Epub 2010 Apr 13. PMID 20392530